CLINICAL TRIAL: NCT02080585
Title: Effectiveness of a Web-based, Computer-tailored, Pedometer-based Physical Activity Intervention for Adults: a Cluster-randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2005/027
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Inactivity
Keywords: Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group without advice (No Intervention): Control group receives no intervention or physical activity advice.
- Computer-tailored physical activity advice (Experimental): Subjects receive computer-tailored physical activity advice.
  Interventions: Behavioral: Physical Activity advice.

INTERVENTIONS:
Behavioral: Physical Activity advice. — Subjects receive advice regarding physical activities.
  Arms: Computer-tailored physical activity advice

SUMMARY:
The present study used a cluster-randomized controlled trial to evaluate the effects of a computer-tailored, pedometer-based Physical Activity (PA) intervention delivered through the Internet. An invitation e-mail with study information was sent to managers of 18 white-collar workplaces. Eight workplaces consented to participate. All employees of a single workplace were allocated at random to either the intervention or a waiting list control group, in order to avoid contamination between employees receiving the intervention and those who were not receiving the intervention. Subsequently, employees of the participating workplaces were recruited by e-mail. Only Dutch speaking employees between 18 and 65 years old, who had access to the Internet at work or at home, were eligible. Interested employees could sign up by returning a confirmation e-mail to the researchers. On receiving this information, a meeting was organized in each of the eight worksites to deliver all documents for baseline measurement (T0) to the participants, including an informed consent form, a blinded pedometer, an activity log and a self-administered questionnaire. During this meeting, information was provided on how to use the pedometer, how to log PA activities and how to answer the questionnaire. Moreover, the participants were asked to adhere to their usual PA pattern throughout the baseline measurement. After one week, all measurement tools were collected, and average daily step counts were calculated. At this point, participants in the intervention condition received (1) a booklet with information on how to increase steps, (2) a non-blinded pedometer, which they could use for three months, and (3) a username, a password and the amount of average daily steps, calculated by the researchers, so that participants could use this number when requesting the online computer-tailored step advice. Participants in the control condition did not receive any of the above mentioned intervention components. One and three months later, all participants again received a blinded pedometer, which was worn for one week. When wearing the blinded-pedometer one month (T1) and three months (T2) post baseline, intervention participants were allowed to also were the non-blinded pedometer. Furthermore, the same self-reported questionnaire was used to measure PA level at T1 and T2 in order to test the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking
* Age range: 18 - 65 years old
* Access to the Internet at work or at home

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Amount of physical activity at baseline. | at baseline
  Using International Physical Activity Questionnaire (IPAQ) and Omron HJ-203-ED pedometer.
Amount of Physical activity 1 month after baseline. | 1 month after baseline
  Using International Physical Activity Questionnaire (IPAQ) and Omron HJ-203-ED pedometer.
Amount of physical activity 3 months after baseline. | 3 months after baseline
  Using International Physical Activity Questionnaire (IPAQ) and Omron HJ-203-ED pedometer.

SECONDARY OUTCOMES:
Sedentary behaviour at baseline. | at baseline
  International Physical Activity Questionnaire (IPAQ)
Sedentary behaviour 1 month after baseline. | 1 month after baseline
  International Physical Activity Questionnaire (IPAQ)
Sedentary behaviour 3 months after baseline. | 3 months after baseline
  International Physical Activity Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Ilse De Bourdeaudhuij, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University - Department of Movement and Sports Sciences, Ghent, Belgium

REFERENCES:
- [Derived] Compernolle S, Vandelanotte C, Cardon G, De Bourdeaudhuij I, De Cocker K. Effectiveness of a web-based, computer-tailored, pedometer-based physical activity intervention for adults: a cluster randomized controlled trial. J Med Internet Res. 2015 Feb 9;17(2):e38. doi: 10.2196/jmir.3402. PMID 25665498